CLINICAL TRIAL: NCT00533637
Title: A Double-Blind, Randomized, Placebo-Controlled, Cross-Over, Allergen Challenge Study to Evaluate Taste and Local Tolerance of NLA Nasal Spray in Patients With Allergic Rhinitis
Brief Title: Taste and Local Tolerance Study of NLA Nasal Spray in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biolipox AB (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLA-C004P
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2007-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Nasal spray; Anti-histamine; Tolerability
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NLA Nasal Spray
  Interventions: Drug: Cetirizine dihydrochloride (10 mg/ml) liposomal formulation
- 2 (Active Comparator)
  Interventions: Drug: Cetirizine dihydrochloride (10 mg/ml) buffer solution
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetirizine dihydrochloride (10 mg/ml) liposomal formulation — 2x110μL in each nostril twice daily for 7 days
  Arms: 1
Drug: Cetirizine dihydrochloride (10 mg/ml) buffer solution — 2x110μL in each nostril, as a single dose
  Arms: 2
Drug: Placebo — Citrate buffer with preservatives
  Arms: 3

SUMMARY:
Evaluation of NLA Nasal Spray with regard to taste perversion and local tolerance

DETAILED DESCRIPTION:
Oral or intranasal antihistamines is the first line treatment for allergic rhinitis. Cetirizine is a second-generation selective antihistamine widely used in an oral formulation for the treatment of allergic rhinitis. Local administration of cetirizine has been shown to reduce symptoms after allergen challenge, and has the potential to shorten the time to onset and decrease systemic side effects. However, local irritation and nasal burning/pain has been reported after nasal administration. For the compliance of the patients taking a nasal spray, the taste and tolerance of the product is of particular importance. NLA Nasal Spray contains cetirizine in a liposomal formulation aiming to improve the tolerability. The present study aims to compare the NLA Nasal Spray with cetirizine in an aqueous formulation and placebo with regard to taste perversion and local tolerance. This will be investigated off-season in patients with seasonal allergic rhinitis after provocation with allergen.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age (inclusive)
* Body Mass Index (BMI) between 18 and 28 kg/m2
* History of pollen-induced seasonal allergic rhinitis for at least two years and otherwise healthy
* Elevated specific IgE to at least one aero allergen or at least one positive skin pick test (SPT)
* Seasonal allergic rhinitis with symptoms provoked by the allergen with a corresponding elevated specific IgE or positive SPT
* Signed written Informed Consent

Exclusion Criteria:

* Perennial allergic rhinitis except for cat and/or dog sensitivity under the condition that these patients are not exposed to cats and dogs
* Soy bean allergy
* Peanut allergy
* Smoking during the last month before study inclusion
* Any upper respiratory tract infection during the period of 2 weeks before the start of the study
* Chronic medication
* Any medication, including herbal medicines, during their last five half-lives (t½)
* Nasal anatomical deviations
* Extensive use of nasal sprays as judged by the Investigator
* Ongoing nasal symptoms as judged by the Investigator
* Known hypersensitivity to cetirizine
* Pregnant or breast-feeding women
* Fertile women not using reliable methods of contraception (i.e. IUD, barrier method, hormonal contraceptives, abstinence)
* Participation in any other investigational study in the last three months
* Inability to adhere to the study plan
* Previous inclusion in this study
* Blood donation during the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Taste perversion scores | 7 days
Local tolerance scores | 7 days

SECONDARY OUTCOMES:
Treatment efficacy | 1 days
Type and incidence of AEs | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Greiff, MD, PhD, Principal Investigator — University of Lund
Locations (1):
- Department of Otorhinolaryngology, Lund University Hospital, Lund, Sweden